CLINICAL TRIAL: NCT04631484
Title: International, Multicenter, Randomized, Single Blind, Placebo-controlled Study of Efficacy and Safety of CITOFLAVIN® in the Acute Period of Head Injury in Adults
Brief Title: International Trial of Efficacy of Cytoflavin in Head Trauma
Acronym: MITRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTF-III-CCT-2019
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Head Trauma,Closed
Keywords: closed head injury; brain concussion; traumatic brain injury; TBI; Craniocerebral Trauma; posttraumatic amnesia
MeSH Terms: conditions — Head Injuries, Closed; Brain Concussion; Brain Injuries, Traumatic; Craniocerebral Trauma | interventions — cytoflavin; Inosine; Niacinamide; Riboflavin; Succinic Acid

STUDY DESIGN:
Intervention Model Description: International, multicenter, randomized, single blind, third party (outcome assessor) blinding
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytoflavin ((Inosine + Nicotinamide + Riboflavin + Succinic Acid) (Experimental): Patients will receive treatment with the study drug, 20 ml twice a day IV, dissolved in 200 ml of 0.9% NS, for 10 days;patients will stay in the hospital for the the entire period of therapy. Observation of patients and assessment of the main parameters of the efficacy and safety will continue for 14 days.
  Interventions: Drug: Cytoflavin ((Inosine + Nicotinamide + Riboflavin + Succinic Acid)
- Placebo (Placebo Comparator): Patients will receive 20 ml placebo (0.9% sodium chloride solution) twice a day IV, dissolved in 200 ml of 0.9% NS, for 10 days; patients will stay in the hospital for the the entire period of therapy. Observation of patients and assessment of the main parameters of the efficacy and safety will continue for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cytoflavin ((Inosine + Nicotinamide + Riboflavin + Succinic Acid) — 20 ml (2 ampoules, 10 ml each) dissolved in 200 ml of 0.9% sodium chloride, intravenously 2 times a day with an interval of 12 ± 2 hours, for 10 days.
  Arms: Cytoflavin ((Inosine + Nicotinamide + Riboflavin + Succinic Acid)
Drug: Placebo — 20 ml of 0.9% sodium chloride (2 ampoules of 10 ml each), added to 200 ml of 0.9% sodium chloride, intravenously 2 times a day with an interval of 12 ± 2 hours, for 10 days
  Arms: Placebo

SUMMARY:
The study will access the efficacy and safety of treatment with CITOFLAVIN® in patients with non-penetrating moderately severe traumatic brain injury (TBI). The study recruits patients 18-60 years with TBI, corresponding to the clinical diagnosis of brain contusion, with GCS score 9 -14 at the time of inclusion , with the estimated time of initiation of therapy within 24 hours from the estimated or established time of trauma, with post-traumatic amnesia, confusion or disorientation and absence of indications for neurosurgery or other surgical intervention under general anesthesia.

Cytoflavin® (Inosine + Nicotinamide + Riboflavin + Succinic Acid) is a combination drug, which improves cerebral blood flow, activates metabolic processes in the central nervous system, restores impaired consciousness, promotes regression of neurological symptoms and improvement of cognitive functions of the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-60 (inclusive).
2. Clinical diagnosis of TBI, cerebral contusion of moderate severity without compression.
3. The written consent of the legal representative or the decision of the council to include the patient in the study.
4. Possibility of a full assessment of eye opening, speech and motor response by GCS.
5. GCS at the time of inclusion 9 - 14 (inclusive).
6. Time of initiation of study drug therapy within 24 hours after the estimated or determined time of injury.
7. The presence of post-traumatic amnesia, confusion and disorientation.
8. Absence of indications for neurosurgery or other surgical intervention under general anesthesia.
9. Normal brain CT scan, or the presence of subarachnoid hemorrhage and / or contusion foci of I-III types according to Kornienko and / or limited or diffuse cerebral edema.
10. The expected duration of hospital stay >= 10 days.
11. Absence of a disabling neurological or mental illness, information about the patient's disability prior to injury.
12. Possibility to perform all procedures stipulated by the study protocol

Exclusion Criteria:

1. The need to use the therapy prohibited by the study protocol.
2. Concomitant injury, except for cases of damage to the skeleton, soft tissues, internal organs, which do not require (1) surgical intervention under general anesthesia, and (2) are not an independent indication for hospital treatment.
3. Past / planned surgical intervention for the current episode of trauma under general anesthesia.
4. Penetrating open TBI.
5. Presence of the following lesions on the results of computed tomography (CT) of the brain performed prior to the patient's randomization:

   1. epidural hematoma or subdural hematoma;
   2. evidence of a previous head injury based on CT results;
   3. type IV contusion foci according to Kornienko's classification.
6. Presence of any of the following risk factors for secondary brain injury at any time after TBI: hypoxia (SpO2 <90% based on pulse oximetry results); hypotension (systolic blood pressure <90 mm Hg) or shock;hypothermia (body temperature <35 ° C); clinical signs of respiratory failure, the need for mechanical ventilation.
7. Drug addiction.
8. Alcohol in saliva >=2 ‰ or a previous diagnosis of alcohol dependence.
9. Depression of consciousness, presumably resulting from other reasons (for example, alcohol, drugs, drugs, poisonous substances).
10. The presence of aphasia due to focal brain damage, which prevents communication with the researcher.
11. Status epilepticus at the time of admission to the hospital or condition after an epileptic seizure.
12. Pregnant and lactating women.
13. Availability of information about concomitant chronic disease in the stage of decompensation.
14. Intolerance to the components of CYTOFLAVIN®, anamnestic data on drug allergy to succinic acid, riboflavin, inosine, or nicotinamide.
15. Severe renal or heart failure requiring restriction of the volume of injected fluid.
16. The presence of a condition or disease that, in the opinion of the investigator, jeopardizes the patient's safety if the patient participates in the study, or may interfere with the performance of examination procedures, an objective assessment of the patient's condition, or distort the assessment of the outcome of TBI.
17. Participation in any clinical study less than 3 months before the start of the study.
18. Patients who are employees of the research center and their families.
19. Language barrier.
20. Availability of information that the patient is a stateless person or a citizen of another state

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Galveston Orientation and Amnesia scale | 7 days
  The proportion of patients with regression of post-traumatic amnesia by day 7 of treatment, defined as having a Galveston score of >75 points on 3 consecutive days, up to and including day 7 of treatment.
Glasgow Outcome scale - Extended (GOS-E) | 90 days
  Assessment by GOS-E after 3 months

SECONDARY OUTCOMES:
Glasgow Coma Scale | 14 days
  Daily assessment by GCS for the period up to 14 days of the study
Barthel Index | 14 days
  Assessement of Barthel Activities of daily living Index on day 14 or discharge, whatever earlier

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Savello, Prof, Study Director — S. M. Kirov Military Medical Academy of the Ministry of Defense of the Russian Federation; Taras A Skoromets, Prof, Study Director — National Medical Research Center of Psychiatry and Neurology named after V.M. Bekhterev
Locations (8):
- West Kazakhstan Medical University named after. M. Ospanov, Aktobe, Kazakhstan
- Russia (7):
  - Ivanovskaya Regional Clinical Hospital, Ivanovo
  - City Clinical Hospital No. 67 named after L.A. Vorokhobov, Moscow
  - Research Institute of Emergency Medicine n.a. N.V. Sklifosovsky, Moscow
  - Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko, Nizhny Novgorod
  - City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - Stavropol Regional Clinical Hospital, Stavropol
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "Central City Clinical Hospital No. 23", Yekaterinburg

REFERENCES:
- [Derived] Kharitonova T, Bragina T, Ivanova E, Savello A, Skoromets T, Petrikov S. A multicenter, international, randomized, single-blind, placebo-controlled study of the efficacy and safety of inosine-nicotinamide-riboflavin-succinic acid in the acute period of traumatic brain injury in adults. Front Neurol. 2026 Jan 2;16:1683976. doi: 10.3389/fneur.2025.1683976. eCollection 2025. PMID 41551305